CLINICAL TRIAL: NCT02740504
Title: A Test of the Spot Respiration Rate Accuracy of the New Reassure Device on Human Subjects
Brief Title: Reassure Spot Respiration Rate Accuracy Compared to SOMNOScreen
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: D22105-106
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Accuracy of Measurement of Respiration Rate
Keywords: Respiration rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects: All 20 subjects. Selected to have a range of ages (18 to less than 75) and BMI from 18.5 to 45

SUMMARY:
A trial conducted within the company with a new non-contact respiration rate (RR) sensor. The device was compared for accuracy in RR measurement with a cleared device, the SOMNOScreen Easy, which uses chest effort bands.

The RR was measured over a short duration on subjects sitting upright in a chair, with the non-contact sensor at various distances from the subject. A total of 20 subjects were tested, from both genders, selected to represent a wide range of age and body mass index

DETAILED DESCRIPTION:
The Reassure uses Radio Frequency (RF) waves to detect the small movements of the human body due to respiration. The reference device, the SOMNOScreen, uses chest effort bands. The Reassure is non-contact and so more comfortable and convenient for quick RR measurement, in a similar way that an Infra-Red thermometer is compared to a traditional under-the-tongue mercury thermometer.

The aim is to explore the variations in the human body that could have an effect on the radio reflection from the human torso, and thus affect the potential detection and accuracy of breathing rate. Factors that could affect non-contact RF performance are:

* High Body Mass Index (BMI) could potentially reduce the chest wall movement during breathing, or alter the nature of the breathing.
* Elderly, thin skin (ie pensioner with low BMI) may have less RF reflection.
* Female breast tissue may have an effect on detection or accuracy.

This was tested at a number of distances from the non-contact sensor and also with the subject having a thick comforter (duvet) laid across them.

The test conditions were

* Distances of 0.5 m, 1.0m and 1.5m between the subject and the RF sensor.
* Additional test condition of comforter (duvet) on the subject when the distance from subject to sensor is 1.0 m.
* Each test condition carried out twice.

The use of the comforter in one test condition is to confirm that the RR measurement by the Reassure is unaffected by the thickness of clothing or blankets being worn.

ELIGIBILITY:
Inclusion Criteria:

* Greater or equal to 18 years old and less than or equal to 75 years old
* BMI within the range of greater or equal to 18 and less than or equal to 45

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 persons selected to cover the range of age and BMI of 18 to 45
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Phillips, MA, MSc, Principal Investigator — ResMed Sensor Technologies

IPD SHARING:
Plan to Share IPD: No
Trial is for device performance validation and only recorded with Clinical Trials.gov as it involved human volunteers. No intent to publish

REFERENCES:
- [Background] Lim WS, Carty SM, Macfarlane JT, Anthony RE, Christian J, Dakin KS, Dennis PM. Respiratory rate measurement in adults--how reliable is it? Respir Med. 2002 Jan;96(1):31-3. doi: 10.1053/rmed.2001.1203. PMID 11863207

RESULTS

PARTICIPANT FLOW:
Groups:
- Respiration Rate Sensor: All 20 subjects. Selected to have a range of ages (18 to 75) and BMI from 18.5 to 45.
  Actual:
  Age 18 to 30 - quantity 12 31 to 49 - quantity 5 50 to 65 - quantity 3 BMI 18.5 to 24.9 (normal) - quantity 8 25 to 29.9 (overweight) - quantity 9 30 to 45 (obese) - quantity 3
Period: Overall Study
Arm/Group | Respiration Rate Sensor
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Respiration Rate Sensor: All 20 subjects. Selected to have a range of ages (18 to less than 75) and BMI from 18.5 to 45
Arm/Group | Respiration Rate Sensor
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  Ireland | 20

OUTCOME MEASURES:

1. Primary Outcome: Respiration Rate Accuracy
Description: The respiration rate measured contemporaneously by the Reassure and the reference device, SomnoScreen, are compared on a second-by-second basis, over the recording duration. The difference between the two respiration rate measurements (the delta) for all 20 subjects' recordings, in all positions, are plotted on a normal distribution chart, giving 8,800 data points. The distribution chart reveals the mean difference between the two devices' measurements and the Standard Deviation (SD). The measure of success is if the 95% (ie 2SD) of the difference in the respiration rate indicated by the two devices (the delta) is less than 5 breaths per minute. This measure is derived from the peer review paper by Lim et al, cited in the References section
Time Frame: Recording duration of 2 minutes; measurement made after 45 seconds settling time, for at least 60 seconds
Measure: Mean (Standard Deviation); unit: breaths per minute
Groups:
- Respiration Rate Sensor: All 20 subjects. Selected to have a range of ages (18 to less than 75) and BMI from 18.5 to 45.
  Actual:
  Age 18 to 30 - quantity 12 31 to 49 - quantity 5 50 to 65 - quantity 3 BMI 18.5 to 24.9 (normal) - quantity 8 25 to 29.9 (overweight) - quantity 9 30 to 45 (obese) - quantity 3
Arm/Group | Respiration Rate Sensor
Number analyzed (Participants) | 20
breaths per minute | 0.4 (1.75)

ADVERSE EVENTS:
Arm/Group | Respiration Rate Sensor
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes